CLINICAL TRIAL: NCT02932150
Title: A Randomized, Double-Blind Evaluation of the Pharmacokinetics, Safety, and Antiviral Efficacy of Tenofovir Alafenamide (TAF) in Children and Adolescent Subjects With Chronic Hepatitis B Virus Infection
Brief Title: Study of Tenofovir Alafenamide (TAF) in Children and Teen Participants With Chronic Hepatitis B Virus Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-320-1092; 2016-000785-37 (EudraCT Number); 2023-506143-42 (Other: European Medicines Agency)
Record Dates: First submitted 2016-09-16; First posted 2016-10-13 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B
Keywords: CHB; HBV
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- TAF (Cohort 1) (Experimental): Participants (12 to < 18 years) weighing ≥ 35 kg will receive TAF 25 mg tablet for 24 weeks
  Interventions: Drug: TAF
- Placebo (Cohort 1) (Placebo Comparator): Participants (12 to < 18 years) weighing ≥ 35 kg will receive placebo tablet for 24 weeks
  Interventions: Drug: Placebo
- TAF (Cohort 2 Group 1) (Experimental): Participants (6 to < 12 years) weighing ≥ 25 kg will receive TAF 25 mg tablet for 24 weeks
  Interventions: Drug: TAF
- TAF (Cohort 2 Group 2) (Experimental): Participants (6 to < 12 years) weighing ≥ 14 kg to < 25 kg will receive TAF 15 mg oral granules for 24 weeks
  Interventions: Drug: TAF
- TAF (Cohort 2 Group 3) (Experimental): Participants (2 to < 6 years) will receive TAF for 24 weeks as follows:
  * weight ≥ 10 kg to < 14 kg (7.5 mg oral granules)
  * weight ≥ 14 kg to < 25 kg (15 mg oral granules)
  The study has reopened and recruitment is initiated only for this cohort for ≥ 10 to < 14 kg at this time.
  Interventions: Drug: TAF
- Cohort 2 Placebo (Placebo Comparator): Participants will receive matching placebo of TAF (tablet or oral granules) for 24 weeks.
  Interventions: Drug: Placebo
- Open-Label TAF (Experimental): Following 24 weeks of blinded randomized treatment, participants will be eligible to participate in an open-label extension phase to receive TAF for an additional 216 weeks.
  Interventions: Drug: TAF

INTERVENTIONS:
Drug: TAF — Administered orally once daily
  Arms: Open-Label TAF; TAF (Cohort 1); TAF (Cohort 2 Group 1); TAF (Cohort 2 Group 2); TAF (Cohort 2 Group 3)
Drug: Placebo — Administered orally once daily
  Arms: Cohort 2 Placebo; Placebo (Cohort 1)

SUMMARY:
The goals of this clinical study are to compare the effectiveness, safety and tolerability of study drug, tenofovir alafenamide (TAF), versus placebo in teens and children with CHB and to learn more about the dosing levels in children.

ELIGIBILITY:
Key Inclusion criteria:

* Males and non-pregnant, non-lactating females
* Weight at screening as follows:

  * Cohort 1 = ≥ 35 kg (≥ 77 lbs)
  * Cohort 2 Group 1 = ≥ 25 kg (≥ 55 lbs)
  * Cohort 2 Group 2 = ≥ 14 kg to < 25 kg (≥ 30 lbs to <55 lbs)
  * Cohort 2 Group 3 = ≥ 10 kg to < 14 kg (≥ 22 lbs to < 30 lbs) or

    * 14 kg to < 25 kg (≥ 30 lbs to < 55 lbs)
* Willing and able to provide written informed consent/assent (child and parent/legal guardian)
* Documented evidence of CHB (eg, HBsAg-positive for ≥ 6 months)
* HBeAg-positive, or HBeAg-negative, chronic HBV infection with all of the following:

  * Screening HBV DNA ≥ 2 × 10^4 IU/mL
  * Screening serum ALT > 45 U/L (> 1.5 × ULN: 30 U/L) and ≤ 10 × ULN (by central laboratory range)
* Treatment-naive or treatment-experienced will be eligible for enrollment.
* Estimated creatinine clearance (CLCr) ≥ 80 mL/min/1.73m^2 (using the Schwartz formula)
* Normal ECG

Key Exclusion criteria:

* Females who are pregnant or breastfeeding
* Males and females of reproductive potential who are unwilling to use an "effective", protocol-specified method(s) of contraception during the study.
* Coinfection with hepatitis C virus (HCV), HIV, or hepatitis D virus (HDV)
* Evidence of hepatocellular carcinoma (Note: if screening alpha-fetoprotein (AFP) is < 50 ng/mL no imaging study is needed; however, if the screening AFP is > 50 ng/mL an imaging study is required)
* Any history of, or current evidence of, clinical hepatic decompensation
* Abnormal hematological and biochemical parameters
* Chronic liver disease of non-HBV etiology (e.g., hemochromatosis, alpha-1 antitrypsin deficiency, cholangitis)
* Received solid organ or bone marrow transplant
* Currently receiving therapy with immunomodulators (eg, corticosteroids), or immunosuppressants
* Significant renal, cardiovascular, pulmonary, or neurological disease in the opinion of the Investigator
* Malignancy within the 5 years prior to screening. Individuals under evaluation for possible malignancy are not eligible.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with subject compliance.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Serious Adverse Events (SAEs) at Week 24 | Week 24
Incidence of Treatment-Emergent Adverse Events (AEs) at Week 24 | Week 24
Percentage of participants with plasma HBV DNA < 20 IU/mL at Week 24 | Week 24
PK Parameter: AUCtau of TAF for participants from Cohort 2 Part A | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 or 12
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).

SECONDARY OUTCOMES:
Percentage of participants experiencing graded laboratory abnormalities | Weeks 24, 48, 96, and 240
Development as measured by Tanner Stage Assessment | Weeks 24, 48, 96, and 240
Percentage change from baseline in bone mineral density (BMD) of whole body (minus head) by dual imaging x-ray absorptiometry (DXA) | Baseline; Weeks 24, 48, 96, and 240
Percentage change from baseline in BMD of lumbar spine by DXA | Baseline; Weeks 24, 48, 96, and 240
Change from baseline in serum creatinine | Baseline; Weeks 4, 8, 12, 24, 48, 96, and 240
Change from baseline in estimated glomerular filtration rate (eGFR) by the Schwartz formula | Baseline; Weeks 24, 48, 96, and 240
Incidence of treatment-emergent SAEs in participants treated with TAF or placebo for 24 weeks followed by open-label TAF at Weeks 48, 96 and 240 | Weeks 48, 96, and 240
Incidence of treatment-emergentAEs in participants treated with TAF or placebo for 24 weeks followed by open-label TAF at Weeks 48, 96 and 240 | Weeks 48, 96, and 240
Change from baseline in retinol-binding protein to creatine ratio at Weeks 4, 8, 12, 24, and 48 | Baseline; Weeks 4, 8, 12, 24, and 48
Change from baseline in beta-2-microglobulin to creatine ratio at Weeks 4, 8, 12, 24, and 48 | Baseline; Weeks 4, 8, 12, 24, and 48
Change from baseline in glucose at Weeks 4, 8, 12, 24, and 48 | Baseline; Weeks 4, 8, 12, 24, and 48
Change from baseline in phosphate at Weeks 4, 8, 12, 24, and 48 | Baseline; Weeks 4, 8, 12, 24, and 48
Percentage of participants with plasma HBV DNA < 20 IU/mL at Weeks 48, 96, and 240 | Weeks 48, 96, and 240
Proportion of participants with plasma HBV DNA < 20 IU/mL (target not detected) at Weeks 24, 48, 96, and 240 | Weeks 24, 48, 96, and 240
Percentage of participants with alanine aminotransferase (ALT) normalization at Weeks 24, 48, 96, and 240 | Weeks 24, 48, 96, and 240
Composite endpoint of percentage of participants with ALT normalization and HBV DNA < 20 IU/mL at Weeks 24, 48, 96 and 240 | Weeks 24, 48, 96 and 240
Change from baseline in fibrosis as assessed by FibroTest at Weeks 24, 48, 96, and 240 | Baseline; Weeks 24, 48, 96, and 240
Percentage of participants with hepatitis B e antigen (HBeAg) loss and seroconversion to anti-HBe (HBeAG-positive participants only) at Weeks 24, 48, 96, and 240 | Weeks 24, 48, 96, and 240
Percentage of participants with composite endpoint of HBeAg seroconversion and HBV DNA < 20 IU/mL at Weeks 24, 48, 96, and 240 (in HBeAg-positive participants only) | Weeks 24, 48, 96, and 240
Percentage of participants with composite endpoint of ALT normalization, HBeAg seroconversion and HBV DNA < 20 IU/mL at Weeks 24, 48, 96, and 240 (in HBeAg-positive participants only) | Weeks 24, 48, 96, and 240
Percentage of participants with hepatitis B surface antigen (HBsAg) loss and seroconversion to anti-HBs at Weeks 24, 48, 96, and 240 | Weeks 24, 48, 96, and 240
Percentage of participants with qHBsAg log10 IU/mL at Weeks 24, 48, 96, and 240 | Weeks 24, 48, 96, and 240
Incidence of resistance mutations at Weeks 24, 48, 96, and 240 | Weeks 24, 48, 96, and 240
Acceptability of study drug | Baseline; Weeks 4, 24, and 36
  To assess acceptability of study drug, the investigator will ask participants if they were able to taste the medication on a scale of 1-5, how much they like the taste of the medication (1 = dislike very much to 5 = like very much).
Palatability of study drug | Baseline; Weeks 4, 24, and 36
  To assess palatability of study drug, the investigator will ask participants on a scale of 0-3 how easy it was to swallow the pill (0 = poor to 3 = excellent).
PK Parameter: AUCtau of tenofovir (TFV) | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
PK Parameter: AUClast of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
PK Parameter: Ctau of TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  Ctau is defined as the observed drug concentration at the end of the dosing interval.
PK Parameter: Cmax of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: Clast of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  Clast is defined as the last observable concentration of drug.
PK Parameter: Tmax of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  Tmax is defined as the time of Cmax (the maximum concentration of drug).
PK Parameter: Tlast of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  Tlast is defined as the time (observed time point) of Clast.
PK Parameter: λz of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug.
PK Parameter: CL/F of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  CL/F is defined as the apparent oral clearance following administration of the drug.
PK Parameter: Vz/F of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  Vz/F is defined as the apparent volume of distribution of the drug.
PK Parameter: t1/2 of TAF and TFV | Predose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, and 8 hours postdose at Week 4 or 8 (Cohort 1), and Week 4, 8, or 12 (Cohort 2)
  t1/2 is defined as the estimate of the terminal elimination half-life of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (62):
- United States (22):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Rady Childrens Hospital, San Diego, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Miami/Schiff Center for Liver Diseases, Miami, Florida
  - AdventHealth Medical Group, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital - Main Hospital, Houston, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
- Cliniques Universitaires Saint-LUC UCL, Brussels, Belgium
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - BC Children's Hospital, Vancouver
- Prince of Wales Hospital, Shatin, Hong Kong
- India (13):
  - GCS Medical Hospital & Research Center, Ahmedabad
  - SR Kalla Memorial Gastro And General Hospital, Jaipur
  - Pratha Gastro Liver Center, Kanpur
  - Institute of Post Graduation Medical Education & Research, Kolkata
  - M. V Hospital and Research Center, Lucknow
  - Seth GS Medical College and KEM Hospital, Mumbai
  - LTMMC & LTMG Hospital, Mumbai
  - Nandita Hospital and Research Centre, Nagpur
  - Khalatkar Hospital, Nagpur
  - Midas Multispecility Hospital PVT. LTD., Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - SIDS Hospital and Research Centre, Surat
  - Samvedna Hospital, Varanasi
- AOU di Bologna - Policlinico S. Orsola Malpighi - Dipartimento Malattic dell'Apparato Digerente e Medicina Intema, Bologna, Italy
- Auckland Clinical Studies Limited, Auckland, New Zealand
- Romania (2):
  - Spitalul Grigore Alexandrescu-Sectia Pediatrie III, Bucharest
  - Institutul National de Boli Infectioase "Prof.Dr. Matei Bals", Bucharest
- Russia (8):
  - Krasnoyarsk Regional Clinical Center of Maternal and Child Welfare, Krasnoyarsk
  - Federal Budgetary Institution of Science "Central Scientific-Research Institute of Epidemiology", Moscow
  - Federal Research Centre of Nutrition, Biotechnology and Food Safety, Moscow
  - Scientific Center of Children's Health of the Ministry of Health of the Russian Federation, Moscow
  - Federal State-Financed Institution Pediatric Research and Clinical Center for Infectious Diseases, Saint Petersburg
  - Federal Budgetary Scientific Institution Pasteur St. Petersburg Scientific Research Institute of Epidemiology and Microbiology, Saint Petersburg
  - Republican Clinical Hospital of Infectious Diseases named after A.F. Agafonov, Tatarstan
  - Limited Medical Company Hepatolog, Tolyatti
- South Korea (5):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Mackay Memorial Hospital, Taipei
  - Chang Gung Medical Foundation, Chang Gung Memorial Hospital, Linkou, Taoyuan District

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-320-1092